CLINICAL TRIAL: NCT03429959
Title: SOCKNLEG Compression Stocking Kit User Friendliness: Donning-Doffing-Edema Prevention An Open Monocentric Randomized Controlled Cross-over Trial
Brief Title: SOCKNLEG Compression Stocking Kit : User Friendliness
Acronym: SOCKNLEGZH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SL1725
Record Dates: First submitted 2017-12-15; First posted 2018-02-12 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Venous Insufficiency of Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOCKNLEG (Experimental): Donning and doffing success of the study stocking compared with both stockings, wearing of the study stocking for a day, standardized non invasive measurement to calculate leg volume of the study leg
  Interventions: Device: SOCKNLEG
- SIGVARIS Cotton (Active Comparator): Donning and doffing success of the study stocking compared with both stockings, wearing of the study stocking for a day, standardized non invasive measurement to calculate leg volume of the study leg
  Interventions: Device: SIGVARIS Cotton

INTERVENTIONS:
Device: SOCKNLEG — Donning and doffing success compared with the two study stockings, wearing the assigned study stocking for a day, Patient Quesationnaire on donning and doffing success and wearing comfort of each study stocking
  Arms: SOCKNLEG
Device: SIGVARIS Cotton — SIGVARIS Cotton
  Arms: SIGVARIS Cotton

SUMMARY:
The investigators aim to evaluate the user friendliness of a newly designed leg compression stocking kit, the SOCKNLEG, compared to a standard leg compression stocking of the same compression strength, the SIGVARIS Cotton. The SOCKNLEG is not yet commercially available, whereas the SIGVARIS Cotton has been successfully commercialized for many years.

After an initial screening visit, a computer generated list will allocate the participants in either the SOCKNLEG or the SIGVARIS Cotton group.

All participants will try on both study stockings, in the order of their allocated group, and will rate their donning and doffing success with a questionnaire. The patients will then wear only the assigned study stocking of their allocated group, for a day and rate its comfort again at the end of the day. The donning and doffing success will also be rated by the study investigator. Leg volume measurements of the study leg will be taken at each visit to determine edema prevention.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Male or postmenopausal female patient, aged over 65 years of age
* Diagnosed venous insufficiency stage C3-C6 (according to CEAP (Clinical, Etiologic, Anatomic, Pathophysiologic) -classification for venous diseases)

Exclusion Criteria:

* Venous leg ulcer with a surface >5cm2
* Peripheral artery disease (PAD) or media calcinosis (Ankle-Brachial-Index <0.8 or >1.3)
* Difference in brachial blood pressure >20mmHg in both arms
* Suspected polyneuropathy with ≥4 sensible test areas, measured with the Semmes-Weinstein-Monofilament-Test
* Inability to reach the forefoot with their hands
* Inability to follow the procedures of the study
* Bed-ridden hospitalized patients who are not able to leave the bed or sit upright for a few consecutive hours

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who completely don the two investigated leg compression devices | through study completion, within 7 months

SECONDARY OUTCOMES:
Number of patients who completely doff the two investigated leg compression devices | through study completion, within 7 months
Patient evaluation of user friendliness | 3 days
  Evaluation of user friendliness using the ICC compression questionnaire
Measuring oedema prevention of the compression stockings by comparison of leg volume measurement at V4 to V3 and V4 to V2. | 3 days
  Assessment by measuring leg volume at the morning visit 3, compared to leg volume at the evening visit 4 and by comparing the leg volumes of visit 4 (compression) to visit 2 (no compression for 1 day)
Time needed to don and doff the two investigated leg compression | 3 days
  Time in minutes and seconds needed to don and doff each study stocking, measured by study investigator

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Hafner, Prof., Principal Investigator — Department of Dermatology, University Hospital Zurich, Zurich, Switzerland
Locations (1):
- Department of Dermatology, University Hospital of Zurich, Switzerland, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No